CLINICAL TRIAL: NCT04294069
Title: Azithromycin Pharmacokinetics and Pharmacodynamics in Pregnancy and Preterm Birth Prevention: Optimizing Dosing to Improve Maternal and Neonatal Outcomes
Brief Title: Azithromycin Dose and PPROM Treatment: a Pilot Randomized Controlled Trial
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20G.119
Record Dates: First submitted 2020-02-18; First posted 2020-03-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin 500mg (Active Comparator): 500mg azithromycin PO daily for seven days
  Interventions: Drug: Azithromycin 500 mg
- Azithromycin 1000mg (Active Comparator): 1000mg azithromycin PO once at admission
  Interventions: Drug: Azithromycin Oral Product

INTERVENTIONS:
Drug: Azithromycin 500 mg — 500mg azithromycin PO for seven days starting on admission
  Arms: Azithromycin 500mg
Drug: Azithromycin Oral Product — 1000mg azithromycin PO once at admission
  Arms: Azithromycin 1000mg

SUMMARY:
This is a pilot randomized controlled trial to assess the pharmacokinetics and pharmacodynamics of azithromycin in pregnant singletons admitted with preterm premature rupture of membranes (PPROM) at 24 0/7- 33 0/7. Participants will be randomized 1:1 to either 1000mg azithromycin orally once or 500mg azithromycin orally daily for seven days in addition to standard care.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial to assess the pharmacokinetics and pharmacodynamics of azithromycin in pregnant singletons admitted with preterm premature rupture of membranes (PPROM) at 24 0/7- 33 0/7. Participants will be randomized 1:1 to either 1000mg azithromycin orally once or 500mg azithromycin orally daily for seven days in addition to standard care. During the course of eight days participants will have serial collection of amniotic fluid, maternal serum; and at delivery, of placenta, membrane, and cord blood. After delivery, neonatal respiratory samples will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation 24 0/7 -33 0/7 weeks'
* Diagnosed with preterm premature rupture of membranes:

  * History consistent with ruptured membranes (ie leaking, gush of fluid)
  * Sterile speculum exam with pooling
  * Fluid positive for ferning and/or nitrazine
  * With or without confirmatory test such as Amnisure

Exclusion Criteria:

* • Contraindication to azithromycin

  * Active labor, abruption, chorioamnionitis at enrollment
  * Other contraindication to expectant management of PPROM at enrollment

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Azithromycin trough in amniotic fluid | 8 days
  Primary outcome is the mean difference in azithromycin trough (Cmin) in amniotic fluid between the two dosing regimens using nonparametric test

SECONDARY OUTCOMES:
IL-6 in amniotic fluid | 8 days
  Mean difference in IL-6 at delivery or 8 days (which ever is first)
IL-8 in cord blood | 3 months (delivery)
  Mean difference in IL-8 in cord blood
Respiratory ureaplasma colonization in neonate | 3 months
  Culture of nasopharyngeal swab within 48 hours of delivery in neonates
Latency to delivery | 3 months
  Number days from admission to delivey
Intra-amniotic infection | 3 months (delivery)
  Incidence of maternal intra-amniotic infection at delivery
Trend in amniotic fluid cytokines | 8 days
  TNF alpha, IL-1B, IL-6, IL-8 over 8 day period from admission
ureaplasma colonization of membranes | 3 months
  Culture swab taken of membranes after delivery
Histologic chorioamnionitis | 3 months (delivery)
  incidence of histologic chorioamnionitis in placental pathology

CONTACTS AND LOCATIONS:
Overall Officials: Rupsa C Boelig, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD available on request pending completion of data sharing agreement and approval of information requested
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after publication of results
Access Criteria: IPD available on request pending completion of data sharing agreement and approval of information requested